CLINICAL TRIAL: NCT05144997
Title: LORLATINIB (PF-06463922) CONTINUATION PROTOCOL: AN OPEN-LABEL, SINGLE-ARM CONTINUATION STUDY FOR PARTICIPANTS WITH ALK-POSITIVE OR ROS1-POSITIVE NON-SMALL CELL LUNG CANCER (NSCLC) CONTINUING FROM PFIZER SPONSORED LORLATINIB CLINICAL STUDIES
Brief Title: Lorlatinib Continuation Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7461039; 2023-508952-21-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Non-Small-Cell Lung Cancer; NSCLC
Keywords: ALK; anaplastic lymphoma kinase
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lorlatinib (Experimental): Lorlatinib single agent, 100 mg (4 x 25 mg) oral tables, QD, continuously
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — ALK-positive NSCL treatment
  Other Names: PF-06463922

SUMMARY:
The purpose of this protocol is to provide continued treatment access and safety follow-up for eligible participants who continue to derive a benefit from study intervention in the Pfizer sponsored lorlatinib parent studies that will be closed. Additional follow-up safety data collection will permit further characterization of the safety profile of lorlatinib in participants continuing to receive study intervention

ELIGIBILITY:
Inclusion Criteria:

1 - Any participant who is receiving study treatment and deriving clinical benefit (as determined by the Principal Investigator) in a Pfizer-sponsored Lorlatinib Parent Study.

2- Participants must agree to follow the reproductive criteria. 3- Adequate Bone Marrow, Liver, Renal, Pancreatic Function

Exclusion Criteria:

1 - Female participants who are pregnant or breastfeeding. 2- Any medical reason that, in the opinion of the Investigator or Sponsor, precludes the participant from inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events leading to permanent discontinuation of study intervention | Baseline up to approximately 5 years
  Safety collection in this study will permit further characterization of the safety profile of lorlatinib
Number of serious adverse events reported for all participants | Baseline up to approximately 5 years
  Safety collection in this study will permit further characterization of the safety profile of lorlatinib

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California, United States
- China (17):
  - The First affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Hunan Provincial Tumor Hospital, Changsha, Hunan
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The first hospital of jilin university, Changchun, Jilin
  - Sir Run Shaw Hospital, Hangzhou, Qiantang District
  - The Second Affiliated Hospital of PLA Air Force Medical University, Xi'an, Shaanxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer hospital, Chengdu, Sichuan
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - Fudan University Shanghai Cancer Center, Shanghai
- France (2):
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Institut Gustave Roussy, Villejuif
- India (2):
  - Healthcare Global Enterprises, Bengaluru, Karnataka
  - Bhaktivedanta Hospital & Research Institute, Thane, Maharashtra
- Aichi Cancer Center Hospital, Nagoya, Aichi-ken, Japan
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461039